CLINICAL TRIAL: NCT02198820
Title: Practice Survey on Femoral Neck Fractures and the Incidence of Type of Anesthesia on Patient Outcome in the Saint-Luc Bouge Hospital
Brief Title: Practice Survey on Femoral Neck Fractures and the Incidence of Type of Anesthesia on Patient Outcome
Status: Withdrawn | Type: Observational
Why Stopped: lack of investigators
Sponsor: Astes (Other)
Responsible Party: Principal Investigator, Eric DEFLANDRE, MD, FCCP, Eric DEFLANDRE, MD, FCCP, Astes
Other Study IDs: FNF-SLBO
Record Dates: First submitted 2014-07-23; First posted 2014-07-24 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Femoral Neck Fractures
Keywords: Femoral Neck Fractures; Perioperative Care; Perioperative Period; Postoperative Complications
MeSH Terms: conditions — Femoral Neck Fractures; Postoperative Complications | interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- General: All patients included who underwent surgery with general anesthesia
  Interventions: Drug: General Anesthesia
- Loco Regional: All patients included who underwent surgery with loco regional anesthesia
  Interventions: Drug: Loco Regional Anesthesia

INTERVENTIONS:
Drug: General Anesthesia — General anesthesia with proposal, rocuronium and sufentanil
  Groups: General
Drug: Loco Regional Anesthesia — Loco Regional Anesthesia with marcaine
  Groups: Loco Regional

SUMMARY:
Inclusion of all patients with femoral neck fracture presenting in Saint-Luc Bouge Hospital between October 1th 2014 and September 30th 2015.

Comparison of severity scores of these patients and the scale of Nottingham on immediate (day 1 and day 2) and late (1 month) outcome.

DETAILED DESCRIPTION:
Inclusion of all patients with femoral neck fracture presenting in Saint-Luc Bouge Hospital between October 1th 2014 and September 30th 2015.

Comparison of severity scores of these patients and the scale of Nottingham on immediate (day 1 and day 2) and late (1 month) outcome.

This comparison includes preoperative parameters (hemoglobin, creatinine, mini-mental test) and intraoperative parameters (such as type of anesthesia).

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted at the Saint-Luc Bouge Hospital for a femoral neck fractures between 10/01/2014 and 30/09/2014

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted at the Saint-Luc Bouge Hospital for a femoral neck fractures
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Preoperative assessment | 1 month
  Comparison of the impact of preoperative parameters (such as hemoglobin, creatinine, mini-mental test) on patient outcome.

SECONDARY OUTCOMES:
Perioperative assessment | 1 month
  Comparison of the impact of the type of anesthesia (general versus loco regional) on patient outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Eric P DEFLANDRE, MD, FCCP, Principal Investigator — Astes
Locations (1):
- Clinique Saint-Luc de Bouge, Namur, Namur, Belgium